CLINICAL TRIAL: NCT01246986
Title: Phase 2 Study of LY2157299 in Patients With Hepatocellular Carcinoma
Brief Title: A Study of LY2157299 in Participants With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13665; H9H-MC-JBAK (Other: Eli Lilly and Company); 2010-022338-10 (EudraCT Number)
Record Dates: First submitted 2010-11-01; First posted 2010-11-24 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-01

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — LY-2157299; Sorafenib; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part A Cohort 1-160 milligram (mg) LY2157299 (Experimental): Per the protocol, following an interim analysis, the decision was taken to no longer randomize participants to the 160 mg LY2157299 arm. As of May 25,2012, all newly enrolled participants will receive 300 mg LY2157299.
  80 mg LY2157299 given orally twice daily (BID) for 14 days followed by 14 days off (28-day cycle).
  Participants will continue to receive until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: LY2157299
- Part A Cohort 2 - 300 mg LY2157299 (Experimental): 150 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle).
  Participants will continue to receive until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: LY2157299; Drug: Sorafenib
- Part B - 300 mg LY2157299 (Experimental): 150 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle).
  Participants will continue to receive until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: LY2157299
- Part C Cohort 1 - 160 mg LY2157299 + 800 mg Sorafenib (Experimental): 80 mg LY2157299 given orally BID on Days 1 to 14 in combination with 400 mg Sorafenib BID on days 1 to 28 (28-day cycle).
  Participants will continue to receive until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: LY2157299; Drug: Sorafenib
- Part C Cohort 2 - 300 mg LY2157299 + 800 mg Sorafenib (Experimental): 150 mg LY2157299 given orally BID on Days 1 to 14 in combination with 400 mg Sorafenib BID on days 1 to 28 (28-day cycle).
  Participants will continue to receive until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: LY2157299; Drug: Sorafenib
- Part D Cohort 1 - 160 mg LY2157299 + 8 mg/kg Ramucirumab (Experimental): 80 mg LY2157299 given orally BID on days 1 to 14 in combination with ramucirumab 8 mg/kilogram (kg) intravenous (IV) on days 1 and 15 (28-day cycle).
  Participants will continue to receive until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: LY2157299; Drug: Ramucirumab
- Part D Cohort 2 - 300 mg LY2157299 + 8 mg/kg Ramucirumab (Experimental): 150 mg LY2157299 given orally BID on days 1 to 14 in combination with ramucirumab 8 mg/kg IV on days 1 and 15 (28-day cycle).
  Participants will continue to receive until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: LY2157299; Drug: Ramucirumab

INTERVENTIONS:
Drug: LY2157299 — Administered orally
Drug: Sorafenib — Administered orally
  Arms: Part A Cohort 2 - 300 mg LY2157299; Part C Cohort 1 - 160 mg LY2157299 + 800 mg Sorafenib; Part C Cohort 2 - 300 mg LY2157299 + 800 mg Sorafenib
Drug: Ramucirumab — Administered IV
  Other Names: LY30098016
  Arms: Part D Cohort 1 - 160 mg LY2157299 + 8 mg/kg Ramucirumab; Part D Cohort 2 - 300 mg LY2157299 + 8 mg/kg Ramucirumab

SUMMARY:
The purpose of this study is to estimate the median time to progression in participants with hepatocellular carcinoma (HCC) when treated with LY2157299 as monotherapy and in combination with sorafenib or ramucirumab.

DETAILED DESCRIPTION:
The study consists of four Parts: Part A where HCC participants with an increased alpha-fetoprotein (AFP) level will be treated with either 160 milligrams (mg) LY2157299 or 300 mg LY2157299. Part B where HCC participants with a normal AFP level will be treated with 300 mg LY2157299, Part C where treatment-naïve HCC participants will be treated with 160 mg LY2157299 + sorafenib or 300 mg LY2157299 + sorafenib, and Part D where HCC participants will be treated with either 160 mg or 300 mg LY2157299 + ramucirumab.

Participants who continue to receive benefit from treatment at the time that the study is considered completed, may enter the treatment extension period and continue to receive the study treatment. The end of the study is the date of last visit or last scheduled procedure for the last active subject in the study.

ELIGIBILITY:
Inclusion Criteria:

* Have histological evidence of a diagnosis of HCC not amenable to curative surgery
* Part A: Serum alpha fetoprotein greater than or equal to 1.5 Upper Limits of Normal, Part B: Serum alpha fetoprotein less than 1.5 Upper Limits of Normal. Not applicable for Part C or D
* Child-Pugh Stage: A or B7 for Parts A & B, A for Part C, and D
* Have the presence of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). A lesion that has been previously treated by local therapy will qualify as a measurable or evaluable lesion if there was demonstrable progression following locoregional therapy
* Have given written informed consent prior to any study-specific procedures
* Have adequate hematologic, hepatic and renal function
* Have a performance status of equal to or less than 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* For Parts A & B: Have received sorafenib and have progressed or were intolerant to sorafenib or are ineligible for sorafenib treatment. For Part C: not received previous systemic treatment. For Part D: have received sorafenib and have progressed or were intolerant to sorafenib or are ineligible for sorafenib treatment or have not received prior systemic treatment.
* For Parts A, B, and D: have discontinued sorafenib for at least 2 weeks
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug
* Females with childbearing potential must have had a negative serum pregnancy test less than or equal to 7 days prior to the first dose of study drug
* Are able to swallow capsules or tablets

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 28 days from a clinical trial involving an investigational drug or device or not approved use of a drug or device (other than the study drug used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Known HCC with fibro-lamellar or mixed histology
* Presence of clinically relevant ascites
* History of liver transplant requiring increased immunosuppressive therapy. (Participants on maintenance immunosuppressive therapy after liver transplant are eligible for Part A & B)
* Have received more than 1 line of systemic treatment in Parts A, B and D
* Have moderate or severe cardiac disease:

  1. Have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension
  2. Have documented major electrocardiogram (ECG) abnormalities at the investigator's discretion
  3. Have major abnormalities documented by echocardiography with Doppler
  4. Have predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress
* Have serious preexisting medical conditions that, in the opinion of the investigator, that cannot be adequately controlled with appropriate therapy or would preclude participation in this study
* Females who are pregnant or lactating
* Have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless in complete remission and off all therapy for that disease for a minimum of 3 years. At the discretion of the investigator, hormone-refractory prostate cancer participants who are stable on GnRH agonist therapy and breast cancer participants who are stable on antiestrogen therapy may have that treatment continued
* Have active infection that would interfere with the study objectives or influence study compliance
* For Part C, have a known hypersensitivity to sorafenib or its excipients
* For Part D, have a serious illness or medical condition(s), including but not limited to the following:

  1. The participant has undergone major surgery within 28 days prior to randomization or has undergone central venous access device placement within 7 days prior to randomization
  2. The participant has uncontrolled arterial hypertension ≥150 / ≥90 millimeters of mercury (mm Hg) despite standard medical management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2011-03-30 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (10):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of California, San Francisco, San Francisco, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana Univ Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenslopes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards
- France (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clichy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Créteil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saint-Etienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Herblain
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auckland, New Zealand
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Giannelli G, Santoro A, Kelley RK, Gane E, Paradis V, Cleverly A, Smith C, Estrem ST, Man M, Wang S, Lahn MM, Raymond E, Benhadji KA, Faivre S. Biomarkers and overall survival in patients with advanced hepatocellular carcinoma treated with TGF-betaRI inhibitor galunisertib. PLoS One. 2020 Mar 25;15(3):e0222259. doi: 10.1371/journal.pone.0222259. eCollection 2020. PMID 32210440
- [Derived] Addepalli A, Kalyani S, Singh M, Bandyopadhyay D, Mohan KN. CalPen (Calculator of Penetrance), a web-based tool to estimate penetrance in complex genetic disorders. PLoS One. 2020 Jan 29;15(1):e0228156. doi: 10.1371/journal.pone.0228156. eCollection 2020. PMID 31995602
- [Derived] Faivre S, Santoro A, Kelley RK, Gane E, Costentin CE, Gueorguieva I, Smith C, Cleverly A, Lahn MM, Raymond E, Benhadji KA, Giannelli G. Novel transforming growth factor beta receptor I kinase inhibitor galunisertib (LY2157299) in advanced hepatocellular carcinoma. Liver Int. 2019 Aug;39(8):1468-1477. doi: 10.1111/liv.14113. Epub 2019 Jun 3. PMID 30963691
- [Derived] Li S, Yang F, Ren X. Immunotherapy for hepatocellular carcinoma. Drug Discov Ther. 2015 Oct;9(5):363-71. doi: 10.5582/ddt.2015.01054. PMID 26632545
- See also: A Study of LY2157299 in Participants With Hepatocellular Carcinoma — https://www.lillytrialguide.com/en-US/studies/liver-cancer/JBAK#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had progressive disease or death are defined as completed. Per the protocol, following an interim analysis, the decision was taken to no longer randomize participants to the 160 mg LY2157299 arm.
Groups:
- Part A Cohort 1 - 160 mg LY2157299: 80 mg LY2157299 given orally twice daily (BID) for 14 days followed by 14 days off (28-day cycle).
- Part A Cohort 2 - 300 mg LY2157299; Part B - 300 mg LY2157299: 150 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle).
- Part C Cohort 1 - 160 mg LY2157299 + Sorafenib: 80 mg LY2157299 given orally BID on Days 1 to 14 in combination with 400 mg Sorafenib BID on days 1 to 28 (28-day cycle).
- Part C Cohort 2 - 300 mg LY2157299 + Sorafenib: 150 mg LY2157299 given orally BID on Days 1 to 14 in combination with 400 mg Sorafenib BID on days 1 to 28 (28-day cycle).
- Part D Cohort 1 - 160 mg LY2157299 + Ramucirumab: 80 mg LY2157299 given orally BID on days 1 to 14 in combination with ramucirumab 8 mg/kilogram (kg) intravenous (IV) on days 1 and 15 (28-day cycle).
- Part D Cohort 2 - 300 mg LY2157299 + Ramucirumab: 150 mg LY2157299 given twice orally BID on days 1 to 14 in combination with ramucirumab 8 mg/kg IV on days 1 and 15 (28-day cycle).
Period: Overall Study
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib | Part D Cohort 1 - 160 mg LY2157299 + Ramucirumab | Part D Cohort 2 - 300 mg LY2157299 + Ramucirumab
Started | 37 | 72 | 40 | 3 | 44 | 3 | 5
Received at Least 1 Dose of Study Drug | 37 | 72 | 40 | 3 | 44 | 3 | 5
Completed | 34 | 67 | 34 | 3 | 40 | 2 | 5
Not Completed | 3 | 5 | 6 | 0 | 4 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 3 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 3 | 0 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Part A Cohort 1 - 160 mg LY2157299: 80 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle)..
- Part A Cohort 2 - 300 mg LY2157299: 150mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle).
- Part D Cohort 2 - 300 mg LY2157299 + Ramucirumab: 150 mg LY2157299 given twice BID on days 1 to 14 in combination with ramucirumab 8 mg/kg IV on days 1 and 15 (28-day cycle).
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib | Part D Cohort 1 - 160 mg LY2157299 + Ramucirumab | Part D Cohort 2 - 300 mg LY2157299 + Ramucirumab | Total
Number analyzed (Participants) | 37 | 72 | 40 | 3 | 44 | 3 | 5 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.8) | 63.3 (10.8) | 68.1 (9.6) | 70.3 (4.7) | 63.7 (9.8) | 54.0 (11.3) | 63.2 (11.2) | 64.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 4 | 0 | 5 | 0 | 0 | 27
  Male | 32 | 59 | 36 | 3 | 39 | 3 | 5 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 7 | 1 | 0 | 6 | 2 | 4 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 7 | 0 | 0 | 9
  Black or African American | 2 | 3 | 1 | 0 | 2 | 0 | 1 | 9
  White | 34 | 58 | 35 | 2 | 20 | 0 | 0 | 149
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 0 | 9 | 1 | 0 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 2 | 5 | 4 | 0 | 12 | 0 | 0 | 23
  United States | 6 | 12 | 4 | 1 | 10 | 3 | 5 | 41
  Italy | 12 | 15 | 9 | 0 | 4 | 0 | 0 | 40
  Australia | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 5
  France | 12 | 27 | 16 | 0 | 14 | 0 | 0 | 69
  Germany | 4 | 7 | 4 | 2 | 4 | 0 | 0 | 21
  Spain | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 5
Alpha-Fetoprotein [Count of Participants; unit: Participants]
  < 200 nanograms per Liter (µg/L) | 9 | 23 | 28 | 2 | 20 | 1 | 2 | 85
  200 - 400 (µg/L) | 3 | 5 | 0 | 0 | 4 | 0 | 0 | 12
  > 400 (µg/L) | 23 | 43 | 0 | 1 | 16 | 2 | 2 | 87
  Unknown/Not reported | 2 | 1 | 12 | 0 | 4 | 0 | 1 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Relationship of Biomarker Alpha-fetoprotein (AFP) to Overall Survival (OS)
Description: Biomarker response was defined as a > 20% decrease in the biomarker AFP from baseline during 8 weeks of treatment. Data presented is median overall survival of those participants who achieved the defined biomarker response. Participants enrolled in Part A had a baseline AFP level of >1.5 upper limit normal (ULN). Participants enrolled in Part B had baseline AFP level <1.5 ULN.
Time Frame: Baseline, discontinuation from any cause (Up to 83 months)
Population: All participants who received at least one dose of study drug, achieved a >20% reduction in biomarker AFP, and had evaluable post-baseline biomarker data. Due to low enrollment into Part C Cohort - 160 mg reporting group, Kaplan Meier analysis for OS was not conducted in this subgroup. Per protocol, Part D collected safety data only.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part A Cohort 1 - 160 mg LY2157299: 80 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle) for Cohort 1.
- Part B LY2157299; Part C LY2157299: 150 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle).
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B LY2157299 | Part C LY2157299
Number analyzed (Participants) | 8 | 14 | 10 | 27
Months | 19.0 [1.5 to 25.1] | 21.5 [2.9 to 34.2] | 24.2 [3.0 to NA] — Part B 95% Confidence Interval (CI) upper limit non-estimable | 17.9 [12.6 to 32.8]

2. Primary Outcome: Change From Baseline in Relationship of Biomarker Transforming Growth Factor - Beta (TGF-β) to Overall Survival (OS)
Description: Biomarker response was defined as a > 20% decrease in the biomarker TGF-B from baseline. Data presented is median overall survival of those participants who achieved biomarker response.
Time Frame: Baseline,discontinuation from any cause (Up to 83 months)
Population: All participants who received at least one dose of study drug, achieved a >20% reduction in biomarker TGF-β and had evaluable post-baseline biomarker data. Due to low enrollment in Part C Cohort 1 - 160 mg reporting group, Kaplan Meier analysis for OS was not conducted in this subgroup. Per protocol, Part D collected safety data only.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part A Cohort 2 - 300 mg LY2157299: 150 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle) for Cohort 2.
- Part C LY2157299: 150 mg LY2157299 given orally BID for 14 days followed by 14 days 0ff (28-day cycle).
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B LY2157299 | Part C LY2157299
Number analyzed (Participants) | 16 | 34 | 28 | 31
Months | 11.9 [5.4 to 15.6] | 10.1 [4.9 to 15.5] | 21.9 [12.4 to NA] — Part B 95% CI upper limit was non-estimable. | 22.88 [16.2 to 31.8]

3. Primary Outcome: Time to Progression (TTP)
Description: TTP is measured from the date of first dose to the first date of progression of disease based on the investigator review of tumor response using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Progression is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: Randomization to date of first measured progressive disease (Up to 36 Weeks)
Population: All participants who receive at least one dose of study drug. Per protocol, Part D collected safety data only.
Measure: Median (90% Confidence Interval); unit: Weeks
Groups:
- Part C Cohort 1 - 160 mg + Sorafenib: 80 mg LY2157299 given orally BID on Days 1 to 14 in combination with 400 mg Sorafenib
- Part C Cohort 2 - 300 mg LY2157299 + Sorafenib: 150 mg LY2157299 given orally BID on Days 1 to 14 in combination with 400 mg Sorafenib BID on days 1 to 28 (28-day
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib
Number analyzed (Participants) | 37 | 72 | 40 | 3 | 44
Weeks | 12.1 [6.3 to 17.6] | 7.1 [6.3 to 12.7] | 18.0 [10.0 to 24.0] | 36.0 [18.0 to 36.0] | 17.9 [12.1 to 24.0]

4. Secondary Outcome: Population Pharmacokinetics (PK) Mean Population Clearance of Galunisertib
Description: Population mean (between-subject coefficient variance [CV %]) apparent clearance.
Time Frame: Cycle (C) 1: Day (D)1: Predose, 0.5-2 hours(h) Postdose; D14: Predose, 0.5-2, 3-5 h, Postdose; D15 Morning; D22 Morning; Predose C2 and C3 Predose D1
Population: All participants who received at least one dose of study drug, regardless of dose, with evaluable PK data. Per protocol, Part D collected safety data only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Groups:
- LY2157299: LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle).
Arm/Group | LY2157299
Number analyzed (Participants) | 143
Liter per hour (L/hr) | 33.6 (48)

5. Secondary Outcome: Recommended Dose for Phase 3 Hepatocellular Carcinoma (HCC) Trials
Time Frame: Cycle 1 (28 Days)
Population: All participants in Part A and Part B.
Measure: Number; unit: milligrams (mg)
Arm/Group | LY2157299
Number analyzed (Participants) | 74
milligrams (mg) | 300

6. Secondary Outcome: Overall Survival (OS)
Description: OS duration is measured from the date of first dose to the date of death from any cause.
Time Frame: Randomization to date of death from any cause (Up to 83 months)
Population: All participants who received at least one dose of study drug. Per protocol, Part D collected safety data only.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib
Number analyzed (Participants) | 37 | 72 | 40 | 3 | 44
Weeks | 39.1 [24.1 to 52.6] | 29.6 [19.6 to 38.6] | 73.0 [45.4 to 104.7] | 30.3 [28.4 to 70.3] | 89.6 [70.3 to 104.9]

7. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS duration is measure from the date of first dose to the first date of objective progression of disease or death from any cause. Progression is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: Randomization to measured progressive disease or death from any cause (Up to 45 Weeks)
Population: All participants who received at least one dose of study drug. Per protocol, Part D collected safety data only.
Measure: Median (90% Confidence Interval); unit: Weeks
Groups:
- Part B - 300 mg LY2157299: 150 mg LY2157299 given orally 150 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle).
- Part C Cohort 1 - 160 mg LY2157299 + Sorafenib: 80 mg LY2157299 given orally BID on Days 1 to 14 in combination with 400 mg Sorafenib BID on days 1 to 28 (28-day
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib
Number analyzed (Participants) | 37 | 72 | 40 | 3 | 44
Weeks | 12 [6.3 to 12.6] | 6.6 [6.1 to 10.9] | 13.4 [7.4 to 23.3] | 28.4 [6.0 to 36.0] | 28.4 [17.4 to 45.3]

8. Secondary Outcome: Percentage of Participants Achieving an Objective Response (Response Rate)
Description: The percentage of participants who achieved best overall response of either Complete Response (CR) or Partial Response (PR). The overall response rate for each dose with be estimated by dividing the number of confirmed responders by the number of participants who received at least one dose of study drug. Per RECIST v.1.0 criteria CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 millimeter (mm). Tumor-marker results must have normalized. PR is defined as at least 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters.
Time Frame: Randomization to measured progressive disease (Up to 36 Weeks)
Population: All participants who received at least one dose of study drug. Per protocol, Part D collected safety data only.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib
Number analyzed (Participants) | 30 | 46 | 27 | 3 | 44
percentage of participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 3.7 | 0 | 2.3

9. Secondary Outcome: Duration of Tumor Response (DoR)
Description: DoR is measured from the date of the first objective status assessment of a Complete Response (CR) or Partial Response (PR), as determined by RECIST v1.1, to the first date of objective progression of disease or death from any cause. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 millimeter (mm). Tumor-marker results must have normalized. PR is defined as at least 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progression is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: Time of response to measured progressive disease or death from any cause (Up to 84 Weeks)
Population: All participants who received at least one dose of study drug with assessment of CR or PR. Per protocol, Part D collected safety data only.
Measure: Median (90% Confidence Interval); unit: Weeks
Groups:
- Part C Cohort 1 - 160 mg LY2157299 + Sorafenib: 80 mg LY2157299 given orally BID on days 1 to 14 in combination with 400 mg Sorafenib BID on days 1 to 28 (28-day cycle
- Part C Cohort 2 - 300 mg LY2157299 + Sorafenib: 150 mg LY2157299 given orally BID on days 1 to 14 in combination with 400 mg Sorafenib BID on days 1 to 28 (28-day cycle
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib
Number analyzed (Participants) | 0 | 0 | 2 | 0 | 4
Weeks |  |  | 37.6 [25.1 to 50.1] |  | 40.2 [12.1 to 84.1]

10. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is measured from the date of first dose until the date of discontinuation of study treatment due to adverse event, progression of disease, or death from any cause.
Time Frame: Randomization to the date of discontinuation of study treatment due to adverse event, progression of disease, or death from any cause (Up to 75 Weeks)
Population: All participants who received at least one dose of study drug. Per protocol, Part D collected safety data only.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib
Number analyzed (Participants) | 37 | 72 | 40 | 3 | 44
Weeks | 13.4 [8.6 to 18.0] | 9.9 [8.1 to 12.1] | 19.3 [12.1 to 26.3] | 26.3 [19.3 to 54.0] | 49.3 [18.3 to 75.3]

11. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy, Hepatobiliary (FACT-Hep) Sub-scores and Total Score
Description: FACT-Hep consists of 45 items in five subscales (1) physical well-being (PWB) score rage 0 -28; (2) social well-being (SWB) score range 0-28; (3) emotional well-being (EWB) score range 0-24; (4) functional well-being (FWB) score range 0-28; and (5) the hepatobiliary cancer subscale (HCS) Score range 0-72; FACT-Hep score range 1-180, and Trial-Outcome Index (TOI) score range 1-128, to assess health related quality of life in participants with cancer. Higher scores reflect a better health state.
Time Frame: Baseline, Day 1 Cycle 4
Population: All participants with baseline and one post-baseline FACT-Hep Questionnaire in Cycles 2, 3, or 4. Per protocol, Part D collected safety data only.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Part C Cohort 1 - 160mg LY2157299 + Sorafenib: 80 mg LY2157299 given orally BID on days 1 to 14 in combination with ramucirumab 8 mg/kilogram (kg) intravenous (IV) on days 1 and 15 (28-day cycle).
- Part C Cohort 2 - 300 mg LY2157299 + Sorafenib: 150 mg LY2157299 given orally BID on days 1 to 14 in combination with ramucirumab 8 mg/kilogram (kg) intravenous (IV) on days 1 and 15 (28-day cycle).
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib
Number analyzed (Participants) | 30 | 51 | 38 | 3 | 39
units on a scale
  PWB | 0.06 (3.6) | -0.16 (5.0) | 0.04 (3.4) | -1.67 (1.5) | -1.75 (4.4)
  SWB | 0.96 (2.9) | 0.24 (3.4) | 0.37 (4.5) | -1.11 (2.8) | 0.41 (3.6)
  EWB | 0.55 (2.7) | 1.17 (3.9) | 1.13 (4.1) | 2.87 (2.8) | 0.85 (2.5)
  FWB | -0.02 (5.3) | 0.84 (3.6) | 1.20 (4.7) | -1.00 (1.0) | -1.19 (4.6)
  HCS: number analyzed (Participants) | 30 | 50 | 38 | 3 | 39
  HCS | 1.93 (7.6) | 1.40 (7.8) | 0.89 (6.8) | 1.08 (6.0) | -3.79 (7.3)
  FACT-Hep | 2.04 (1.53) | 1.50 (17.5) | 0.58 (18.2) | -0.50 (6.5) | -8.54 (17.0)
  TOI | 1.34 (13.3) | 1.14 (14.6) | 1.17 (12.2) | -1.92 (7.7) | -8.28 (13.7)

12. Secondary Outcome: Time to Worsening (TTW) of Symptoms (FACT-Hep)
Description: Time to worsening of symptoms used minimally important differences to evaluate Physical Well Being (PWB), Functional Well Being (FWB), Hepatocellular Cancer Symptoms (HCS), National Comprehensive Cancer Network (NCCN)/FACT Hepatocellular Symptoms (FHS), Trial-Outcome Index (TOI). PWB time to worsening was defined as participants who had change in a subscale of ≥ 2 point decrease from baseline; FWB time to worsening was defined as participants who had change in a subscale of ≥ 2 point decrease from baseline; HCS time to worsening was defined as participants who had change in a subscale of ≥ 5 point decrease from baseline; FHS time to worsening was defined as participants who had change in a subscale of ≥ 2 point decrease from baseline; TOI time to Worsening was defined as participants who had change in the subscale of ≥ 7 point decrease from baseline.
Time Frame: Baseline to the worsening of symptoms (up to 567 days)
Population: All participants who completed a baseline and one post-baseline FACT-Hep TTW questionnaire. Due to low enrollment in Part C Cohort 1 - 160 mg reporting group, time-to-event analysis for TTW was not conducted for this subgroup. Per protocol, Part D collected safety data only.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Part C Cohort 2 - 300mg LY2157299: 150 mg LY2157299 given orally BID for 14 days followed by 14 days off (28-day cycle).
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 2 - 300mg LY2157299
Number analyzed (Participants) | 30 | 61 | 37 | 40
Days
  PWB | 114.0 [30.0 to NA] — Upper value of CI was non estimable | 113.0 [57.0 to NA] — Upper value of CI was non estimable | 113.0 [58.0 to 170.0] | 30.0 [29.0 to 57.0]
  FWB | 57.0 [30.0 to 86.0] | 88.0 [57.0 to 371.0] | 64.0 [30.0 to 172.0] | 30.0 [29.0 to 58.0]
  HCS | 114.0 [57.0 to NA] — Upper value of CI was non estimable | 113.0 [85.0 to NA] — Upper value of CI was non estimable | 170.0 [57.0 to 567.0] | 31.0 [29.0 to 57.0]
  FHS | 55.0 [29.0 to 86.0] | 57.0 [30.0 to 113.0] | 57.0 [30.0 to 113.0] | 30.0 [29.0 to 30.0]
  TOI | 114.0 [57.0 to NA] — Upper value of CI was non estimable | 113.0 [58.0 to 371.0] | 179.0 [57.0 to 567.0] | 30.0 [29.0 to 31.0]

ADVERSE EVENTS:
Time Frame: Baseline up to 41.5 months
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Part D Cohort 1 - 160 mg LY2157299 + Ramucirumab: 80 mg LY2157299 given orally BID on days 1 to 14 in combination with ramucirumab 8 mg/kg IV on days 1 and 15 (28-day cycle).
- Part D Cohort 2 - 300 mg LY2157299 + Ramucirumab: 150 mg LY2157299 given orally BID on days 1 to 14 in combination with ramucirumab 8 mg/kg IV on days 1 and 15 (28-day cycle).
Arm/Group | Part A Cohort 1 - 160 mg LY2157299 | Part A Cohort 2 - 300 mg LY2157299 | Part B - 300 mg LY2157299 | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib | Part D Cohort 1 - 160 mg LY2157299 + Ramucirumab | Part D Cohort 2 - 300 mg LY2157299 + Ramucirumab
All-Cause Mortality (participants affected / at risk) | 33/37 | 63/72 | 26/40 | 3/3 | 36/44 | 2/3 | 5/5
Serious Adverse Events (participants affected / at risk) | 15/37 | 36/72 | 16/40 | 3/3 | 28/44 | 1/3 | 2/5
Other Adverse Events (participants affected / at risk) | 32/37 | 64/72 | 38/40 | 3/3 | 44/44 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1 - 160 mg LY2157299 (N=37) | Part A Cohort 2 - 300 mg LY2157299 (N=72) | Part B - 300 mg LY2157299 (N=40) | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib (N=3) | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib (N=44) | Part D Cohort 1 - 160 mg LY2157299 + Ramucirumab (N=3) | Part D Cohort 2 - 300 mg LY2157299 + Ramucirumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (16) | 3 (5) | 1 (2) | 6 (9) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic haematoma (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A Cohort 1 - 160 mg LY2157299 (N=37) | Part A Cohort 2 - 300 mg LY2157299 (N=72) | Part B - 300 mg LY2157299 (N=40) | Part C Cohort 1 - 160 mg LY2157299 + Sorafenib (N=3) | Part C Cohort 2 - 300 mg LY2157299 + Sorafenib (N=44) | Part D Cohort 1 - 160 mg LY2157299 + Ramucirumab (N=3) | Part D Cohort 2 - 300 mg LY2157299 + Ramucirumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 9 (22) | 13 (23) | 10 (20) | 1 (4) | 12 (17) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (9) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 3 (9) | 0 (0) | 7 (22) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 2 (2) | 5 (5) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 11 (12) | 8 (10) | 1 (1) | 7 (8) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 7 (10) | 4 (4) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 5 (7) | 8 (8) | 2 (3) | 0 (0) | 6 (8) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 11 (14) | 7 (7) | 0 (0) | 6 (8) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 10 (13) | 11 (15) | 1 (2) | 21 (43) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (11) | 15 (21) | 9 (9) | 1 (2) | 12 (17) | 1 (1) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 12 (17) | 6 (11) | 1 (1) | 5 (11) | 0 (0) | 0 (0)
Asthenia (General disorders) | 5 (6) | 6 (6) | 4 (8) | 0 (0) | 6 (14) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 9 (10) | 14 (17) | 14 (15) | 2 (2) | 11 (16) | 0 (0) | 2 (4)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 5 (6) | 14 (16) | 12 (17) | 0 (0) | 10 (12) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (4) | 6 (8) | 2 (2) | 1 (1) | 5 (13) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (5) | 3 (3) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (7) | 0 (0) | 0 (0)
Post abortion infection (Infections and infestations) | 0/5 (0) | 0/13 (0) | 0/4 (0) | 0/0 (0) | 1/5 (1) | 0/0 (0) | 0/0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/5 (0) | 0/13 (0) | 0/4 (0) | 0/0 (0) | 1/5 (1) | 0/0 (0) | 0/0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/5 (0) | 0/13 (0) | 0/4 (0) | 0/0 (0) | 1/5 (1) | 0/0 (0) | 0/0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (5) | 8 (8) | 10 (17) | 3 (7) | 24 (58) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 7 (8) | 7 (7) | 2 (2) | 10 (15) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3) | 5 (5) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (9) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 5 (7) | 0 (0) | 6 (7) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 10 (11) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (6) | 4 (4) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1/32 (1) | 0/59 (0) | 0/36 (0) | 0 (0) | 2/39 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (10) | 6 (7) | 0 (0) | 5 (5) | 1 (1) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2) | 3 (3) | 0 (0) | 4 (5) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 28 (61) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (9) | 9 (10) | 8 (10) | 1 (1) | 12 (16) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 10 (11) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 8 (10) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Per the protocol, following an interim analysis, the decision was taken to no longer randomize participants to the 160 mg LY2157299 arm.

Per protocol, Part D collected safety data only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT01246986/Prot_000.pdf
  • Statistical Analysis Plan (2013-10-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT01246986/SAP_001.pdf